CLINICAL TRIAL: NCT00563563
Title: An Open-Label Study Assessing the Safety and Efficacy of Naltrexone Sustained Release (SR) in Combination With Bupropion Sustained Release (SR) in Overweight and Obese, Nicotine-Dependent Subjects
Brief Title: A Study of Naltrexone SR/ Bupropion SR in Overweight and Obese Subjects Who Are Nicotine-Dependent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB-401
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Nicotine Dependence; Overweight; Obesity
Keywords: Nicotine-dependence in overweight and obese subjects
MeSH Terms: conditions — Tobacco Use Disorder; Overweight; Obesity | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NB32 (Experimental): Naltrexone SR 32 mg/Bupropion SR 360 mg daily subjects will receive ancillary therapy including counseling on smoking cessation, diet and exercise.
  Interventions: Drug: NB32; Behavioral: Ancillary therapy

INTERVENTIONS:
Drug: NB32 — All subjects are to complete a 4 week titration period at which time subjects will be titrated up to a maintenance level of study drug. Subjects will then take the maintenance dose of study drug for an additional 20 weeks.
  Other Names: Contrave; Naltrexone SR 32 mg/Bupropion SR 360 mg daily
Behavioral: Ancillary therapy — During the study, subjects will receive ancillary therapy including counseling on smoking cessation, diet and exercise.

SUMMARY:
The purpose of this study is to determine whether a combination of naltrexone SR and bupropion SR is safe and effective in the treatment of nicotine-dependence in overweight and obese subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Female and male subjects must be 18 to 65 years of age;
2. Have body mass index (BMI) greater than or equal to 27 and less than or equal to 45kg/m2;
3. Have smoked an average of at least 10 cigarettes/day in the preceding year, with < 3 month total abstinence period;
4. Self-reported level of motivation to stop smoking ≥ 7, on a scale of 1-to-10;
5. At least moderately concerned about gaining weight after quitting smoking
6. Women of child-bearing potential, must be non-lactating and agree to use effective contraception throughout the study period and 30 days after discontinuation of study drug;
7. Able to comply with all required study procedures and schedule;
8. Able to speak and read English;
9. Willing and able to give written informed consent.

Key Exclusion Criteria:

1. Obesity of known endocrine origin
2. Serious medical condition
3. History of drug or alcohol abuse or dependence
4. Use of excluded concomitant medications
5. History of surgical or device (e.g. gastric banding) intervention for obesity;
6. History or predisposition to seizures
7. Pregnant or breast-feeding women or planning to become pregnant during the study period or within 30 days of discontinuing study drug;
8. Planned surgical procedure that can impact the conduct of the study;
9. Use of investigational drug, device or procedure within 30 days prior to Screening;
10. Participation in any previous clinical trial conducted by Orexigen Therapeutics;
11. Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Assess rates of smoking cessation defined by continuous abstinence. | 12 weeks

SECONDARY OUTCOMES:
To assess the percent change from baseline in total body weight during the entire study | Baseline to endpoint
To assess the rates of smoking cessation as measured by expired CO levels <10 ppm | 12 and 24 weeks
To assess the change from baseline in tobacco use from baseline as measured by a tobacco use diary | Baseline to endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Nader Oskooilar, M.D., Ph.D., Principal Investigator — Pharmacology Research Institute
Locations (3):
- United States (3):
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California